CLINICAL TRIAL: NCT06746090
Title: Improvement in Class II Molar Relationship Among Orthodontic Patients Reminded Through Text Message and Phone Call as Compared to No Reminders for Wearing Class II Elastics -A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Rashna Hoshang Sukhia, Principal Investigator, Aga Khan University Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-8830-26873
Record Dates: First submitted 2024-08-26; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Compliance, Patient
Keywords: Class II elastics; reminders; molar relationship
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Masking Description: Subjects will be assigned to one of the three study groups using a computer generated randomization list. There will be no blinding in the study. The recruitment of the patients will be performed by the investigator who will explain the objective, the three arms of the study and the allocation to the participants. Allocation concealment will be carried out using opaque concealed envelopes which will be opened until the use of intervention is to be explained to the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reminders for wearing class II elastics through text message (Experimental): Reminders daily via whatsapp text message.
  Interventions: Behavioral: Reminders
- Reminders for wearing class II elastics through phone call (Experimental): Reminders weekly via phone call.
  Interventions: Behavioral: Reminders
- No reminders for wearing class II elastics (No Intervention): No reminder for wearing elastics.

INTERVENTIONS:
Behavioral: Reminders — Group A(Intervention): Patients who will be reminded daily via whatsapp text message.
  Group B(Intervention): Patients who will be asked through a weekly phone call about elastic wear and then motivated.
  Arms: Reminders for wearing class II elastics through phone call; Reminders for wearing class II elastics through text message

SUMMARY:
The objective of this study is to determine the difference in improvement in class II molar relationship among orthodontic patients reminded daily through text message, weekly through phone call as compared to no reminders for wearing class II elastics.

DETAILED DESCRIPTION:
Compliance is an important factor for better orthodontic treatment outcome. To find the best strategy for promoting better communication between patients and doctors and to increase the patient adherence to treatment especially in the field of oral health. This study will help us to find out the best and effective modality for efficient treatment outcomes and to avoid any side effects which can occur due to un-cooperation of patients in wearing appliances.

SAMPLE SIZE:

Sample size was calculated using the following formula:

By using the findings of Richter et al.16 who reported a mean improvement in compliance with high reward group as (64.6 ± 12.8), high award group (68.2 ± 7.8) and for no reminder group as (71.8 ± 6.2). We will require a minimum sample size of 51 orthodontic patients with 17 patients in group 1(reminded daily via whatsapp text message), 17 in group 2 (patients who will be asked through a weekly phone call about elastic wear and then motivated) and 17 in group 3 (patients who will not be reminded or motivated through social media) with an inflation of 10 % for loss to follow up/non-response rate, to achieve 80% power with atleast 10% change in compliance and 10% or less change in coefficient of variation at two sided 5% level of significance.

Settings: Dental clinics, Aga Khan University Hospital, Karachi (AKUH) Study Design: Randomized open label control trial Allocation: Parallel design with 1:1:1 allocation ratio Duration of Study: January - September2024 Sampling Technique: Non probability purposive sampling Allocation: Random block allocation with a block size of 2, 4 and 6

Randomization, blinding and treatment allocation:

Subjects will be assigned to one of the three study groups using a computer generated randomization list. There will be no blinding in the study. The recruitment of the patients will be performed by the investigator who will explain the objective, the two arms of the study and the allocation to the participants. Allocation concealment will be carried out using opaque concealed envelopes which will be opened until the use of intervention is to be explained to the patient. All the measurements will be recorded by the investigator in mm by using overjet scale.

DATA COLLECTION:

Prior to the initiation of the study, ethical consent will be taken from the institutional Ethical Review Committee for clinical trial. Patients visiting the orthodontic clinic at the Aga Khan University Hospital Karachi will be included in this study. Patients signing an informed consent form will receive detailed information regarding the study. Patient demographics and distance between lower first permanent mandibular molar (mesial to its band) to cusp tip of upper canine will be recorded in a proforma.

Study groups:

The patients will be screened using the inclusion and exclusion criteria by the co-investigator. Patients undergoing their ideal treatment plans including elastic supported mechanics will be included in the study. The treatment plans will be formulated by a team of orthodontic consultants and residents after evaluating complete pre-treatment orthodontic records. Eligible participants will be randomly allocated to one of the three groups.

Group A(Intervention): Patients who will be reminded daily via whatsapp text message.

Group B(Intervention): Patients who will be asked through a weekly phone call about elastic wear and then motivated.

Group C(Control): Patients who will not be reminded or motivated through social media.

Then between 3 - 6 months of elastic wear distance will be measured through an overjet scale keeping it mesial to the band of lower first permanent mandibular molar to cusp tip of upper canine.

All participants will receive routine instructions for oral hygiene maintenance and care of the appliances. The investigator will unseal the envelope from Clinical Trials Unit (CTU), containing information regarding the intervention to be used on the participants based on randomization.

Ethical considerations:

The study will be conducted according to the guidelines of World Medical Association's Declaration of Helsinki and the principles of Good Clinical Practice (GCP). Any subsequent protocol amendments will be submitted to ERC and regulatory authorities for approval. The trial will be conducted in compliance with regulations, and a copy of final study report will be submitted to ERC. Reminder and motivational therapy have no side effects rather it increases patient compliance and leads to better treatment outcomes. Elastics have been shown to be effective methods to improve class II molar relationship in orthodontic patients.

Possible risks or benefits:

There are no reports in literature for any adverse events regarding reminder therapy. Benefits of the current study include finding a more effective way to increase patient compliance which can be implemented in orthodontic patients not only for wearing elastics but also for other removable orthodontic appliances.

Adverse events:

There are no adverse events related to reminder therapy reported in the literature.

Right of refusal to participate and withdrawal:

Participants will be given detailed information regarding the trial preceding their decision to either participate or refuse to participate in the study.

Patient confidentiality, access and storage:

The information provided by the participant will remain confidential. Nobody except the investigators will have access to it. Participant's name and identity will not be disclosed at any time. However, the data may be seen by ERC or any local regulatory body. As per GCP and other guidelines, data will be retained for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 15 - 50 years with permanent dentition.
* Patients undergoing fixed orthodontic treatment and requires class II elastics for correcting molar relationship as a part of their treatment plan.
* All patients who will sign the informed consent form.
* Patients having access to smartphones.

Exclusion Criteria:

* Patients with uncontrolled periodontal disease or pulpitis.
* Presence of any dental/ craniofacial anomaly or syndrome like hemifacial microsomia, Downs syndrome, Treacher Collins syndrome, etc

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Improvement in class II molar relationship by using an overjet scale among orthodontic patients through reminders. | 6 months
  Reminders will be given daily through text message, weekly through phone call as compared to no reminders for wearing class II elastics. An overjet scale consisting of markings in mm will be used to measure the distance from mesial of the band of lower first permanent mandibular molar to cusp tip of upper canine.

CONTACTS AND LOCATIONS:
Overall Officials: Rashna R Hoshang Sukhia, BDS, FCPS, Principal Investigator — Aga Khan University Hospital, Karachi
Locations (1):
- Afeefa Abul Barakaat, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF